CLINICAL TRIAL: NCT03524976
Title: LIQUID - Treatment of Dural Arteriovenous Fistulas With SQUID™ Liquid Embolic Agent, A Non-interventional, Observational, Prospective and Multi-center Study
Brief Title: Treatment of Dural Arteriovenous Fistulas With SQUID™ Liquid Embolic Agent
Acronym: Liquid
Status: Completed | Type: Observational
Sponsor: Dr. Markus Alfred Möhlenbruch (Other)
Collaborators: University Hospital Schleswig-Holstein (Other)
Responsible Party: Sponsor-Investigator, Dr. Markus Alfred Möhlenbruch, Principle Investigator, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Other Study IDs: Liquid
Record Dates: First submitted 2018-03-19; First posted 2018-05-15 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Dural Arteriovenous Fistula
Keywords: endovascular treatment; liquid embolization
MeSH Terms: conditions — Central Nervous System Vascular Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Embolization with Squid: All patients with DAVFs are treated with SQUID™ aiming at complete occlusion of the fistula. Each participating center will include patients with DAVFs in whom the liquid embolic agent SQUID™ is planned to be used consecutively in the study. The
  Interventions: Device: Squid

INTERVENTIONS:
Device: Squid — SQUID™ is injected into the vascular site to be treated, under fluoroscopic control. DMSO dissipates in the blood and causes precipitation of EVOH in which the tantalum powder is trapped. It then forms a consistent spongy embolus.
  This embolus solidifies from the outside inwardly while moving distally in the vessel. The non-adhesive character of the embolus allows slow and controlled injections while leaving in place the microcatheter.
  Other Names: non-adhesive liquid embolic agent

SUMMARY:
The purpose of this study is assessment of safety, efficacy, and short-term outcome of SQUID™ in the embolization of Dural Arteriovenous Fistula

DETAILED DESCRIPTION:
Traditionally, there are two therapeutic options for the treatment of Dural Arteriovenous Fistula (DAVF): (1) the surgical approach consisting of craniotomy and ligation of the vein and (2) the endovascular approach with embolization of shunting zone. Onyx™ (EVOH (Ethylene Vinyl Alcohol) in solution in an organic solvent, DMSO (Dimethyl Sulfoxide), is the main embolic agent used for the endovascular treatment of DAVF. During the occlusion procedure with Onyx™, residual malformed compartments become gradually less visible on x-ray to the operator, due to the high radiopacity of Onyx™, resulting in a potential risk during treatment. Moreover, viscosity is frequently not as low as required to penetrate the shunt.Thus, development a new embolization system with lower radiopacity and lower viscosity to achieve improved occlusion is needed. SQUID™ is a new liquid embolic agent, with variable radiopacity and viscosity. The purpose of this study is assessment of safety, efficacy, and short-term outcome of SQUID™ in the embolization of DAVFs .

ELIGIBILITY:
Inclusion Criteria:

* Dural Arteriovenous Fistula requiring endovascular treatment with a Lariboisiere score between 3 - 5

  * Intended usage of SQUID™
  * The patient agrees with the clinical data collection and medical file access.

Exclusion Criteria:

* DAVF with a Lariboisiere score < 3 • Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with Dural Arteriovenous Fistulas who will be treated with SQUID™ aiming at complete occlusion of the fistula. Each participating center will include patients with DAVFs in whom the liquid embolic agent SQUID™ is planned to be used consecutively in the study. The patient cohort will include patients with DAVFs who had not undergone any previous treatment with an embolic agent whatsoever.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-08-29 (Actual)

PRIMARY OUTCOMES:
Morbidity/Mortality | 90-180 days after treatment
  number of patients with permanent morbidity or mortality
Occlusion rate | 90 -180 days after treatment
  number of patients with complete occlusion of the treated Dural Arteriovenous Fistula

SECONDARY OUTCOMES:
DAVF anatomy | Baseline / day 0-1
  Anatomical description of the Dural Arteriovenous Fistula using Lariboisiere classification
modified Rankin Score | Baseline / day 0-1
  Baseline mRS
Approach | Treatment / day 1
  approach path (vessel)
Feeders | Treatment / day 1
  number of feeders embolized,
Volume of Squid | Treatment / day 1
  volume and concentration of SQUID™ injected at each embolization
Ballons | Treatment / day 1
  Binary: for access to DAVF was a balloon catheter used / no balloon used
Coils | Treatment / day 1
  If complete occlusion was not achieved using Squid: Binary Outcome: use of coils or no use of coils
Other | Treatment / day 1
  If complete occlusion was not achieved using Squid: Binary Outcome: use of other embolization agent / no other agent used
Immediate Aneurysm Occlusion | Treatment / Day 1
  1. 50-99% occlusion
  2. < 50% occlusion
Follow-Up Aneurysm Occlusion | 90-180 days after treatment
  1. 50-99% occlusion
  2. < 50% occlusion
Functional health status | 90-180 days after treatment
  based on modified Rankin Scale

CONTACTS AND LOCATIONS:
Overall Officials: Markus Moehlenbruch, PD Dr., Principal Investigator — University Hospital Heidelberg
Locations (7):
- Germany (7):
  - Klnikum Augsburg, Augsburg
  - Klinische und interventionelle Neuroradiologie Vivantes Klinikum Neukölln, Berlin
  - Charité-Universitätsmedizin Berlin, Berlin
  - University Clinic Bochum, Bochum
  - Alfried Krupp Krankenhaus Rüttenscheid, Essen
  - Klinik für Neuroradiologie Universitätsklinikum Freiburg, Freiburg im Breisgau
  - LMU Klinikum der Universität München, München

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cognard C, Gobin YP, Pierot L, Bailly AL, Houdart E, Casasco A, Chiras J, Merland JJ. Cerebral dural arteriovenous fistulas: clinical and angiographic correlation with a revised classification of venous drainage. Radiology. 1995 Mar;194(3):671-80. doi: 10.1148/radiology.194.3.7862961.
- [Background] Narayanan S. Endovascular management of intracranial dural arteriovenous fistulas. Neurol Clin. 2010 Nov;28(4):899-911. doi: 10.1016/j.ncl.2010.03.013. PMID 20816269
- [Background] Rammos S, Bortolotti C, Lanzino G. Endovascular management of intracranial dural arteriovenous fistulae. Neurosurg Clin N Am. 2014 Jul;25(3):539-49. doi: 10.1016/j.nec.2014.04.010. Epub 2014 Jun 2. PMID 24994089
- [Background] Li C, Yang X, Li Y, Jiang C, Wu Z. Endovascular Treatment of Intracranial Dural Arteriovenous Fistulas Presenting with Intracranial Hemorrhage in 46 Consecutive Patients: With Emphasis on Transarterial Embolization with Onyx. Clin Neuroradiol. 2016 Sep;26(3):301-8. doi: 10.1007/s00062-014-0362-y. Epub 2014 Dec 13. PMID 25501269
- [Background] Cognard C, Januel AC, Silva NA Jr, Tall P. Endovascular treatment of intracranial dural arteriovenous fistulas with cortical venous drainage: new management using Onyx. AJNR Am J Neuroradiol. 2008 Feb;29(2):235-41. doi: 10.3174/ajnr.A0817. Epub 2007 Nov 7. PMID 17989374
- [Background] Chiu AH, Aw G, Wenderoth JD. Double-lumen arterial balloon catheter technique for Onyx embolization of dural arteriovenous fistulas: initial experience. J Neurointerv Surg. 2014 Jun;6(5):400-3. doi: 10.1136/neurintsurg-2013-010768. Epub 2013 Jun 8. PMID 23749795
- [Background] Adamczyk P, Amar AP, Mack WJ, Larsen DW. Recurrence of "cured" dural arteriovenous fistulas after Onyx embolization. Neurosurg Focus. 2012 May;32(5):E12. doi: 10.3171/2012.2.FOCUS1224. PMID 22537121
- [Background] Ambekar S, Gaynor BG, Peterson EC, Elhammady MS. Long-term angiographic results of endovascularly "cured" intracranial dural arteriovenous fistulas. J Neurosurg. 2016 Apr;124(4):1123-7. doi: 10.3171/2015.3.JNS1558. Epub 2015 Sep 25. PMID 26406789
- [Background] Akmangit I, Daglioglu E, Kaya T, Alagoz F, Sahinoglu M, Peker A, Derakshani S, Dede D, Belen D, Arat A. Preliminary experience with squid: a new liquid embolizing agent for AVM, AV fistulas and tumors. Turk Neurosurg. 2014;24(4):565-70. doi: 10.5137/1019-5149.JTN.11179-14.0. PMID 25050683
- [Background] Abud TG, Nguyen A, Saint-Maurice JP, Abud DG, Bresson D, Chiumarulo L, Enesi E, Houdart E. The use of Onyx in different types of intracranial dural arteriovenous fistula. AJNR Am J Neuroradiol. 2011 Dec;32(11):2185-91. doi: 10.3174/ajnr.A2702. Epub 2011 Sep 29. PMID 21960490
- [Background] Chandra RV, Leslie-Mazwi TM, Mehta BP, Yoo AJ, Rabinov JD, Pryor JC, Hirsch JA, Nogueira RG. Transarterial onyx embolization of cranial dural arteriovenous fistulas: long-term follow-up. AJNR Am J Neuroradiol. 2014 Sep;35(9):1793-7. doi: 10.3174/ajnr.A3938. Epub 2014 Apr 17. PMID 24742807
- [Background] Gross BA, Albuquerque FC, Moon K, McDougall CG. Evolution of treatment and a detailed analysis of occlusion, recurrence, and clinical outcomes in an endovascular library of 260 dural arteriovenous fistulas. J Neurosurg. 2017 Jun;126(6):1884-1893. doi: 10.3171/2016.5.JNS16331. Epub 2016 Sep 2. PMID 27588586
- [Background] Gallas S, Drouineau J, Gabrillargues J, Pasco A, Cognard C, Pierot L, Herbreteau D. Feasibility, procedural morbidity and mortality, and long-term follow-up of endovascular treatment of 321 unruptured aneurysms. AJNR Am J Neuroradiol. 2008 Jan;29(1):63-8. doi: 10.3174/ajnr.A0757. Epub 2007 Oct 9. PMID 17925369
- [Background] Hsu YH, Lee CW, Liu HM, Wang YH, Chen YF. Endovascular treatment and computed imaging follow-up of 14 anterior condylar dural arteriovenous fistulas. Interv Neuroradiol. 2014 May-Jun;20(3):368-77. doi: 10.15274/INR-2014-10028. Epub 2014 Jun 17. PMID 24976101
- [Background] Long XA, Karuna T, Zhang X, Luo B, Duan CZ. Onyx 18 embolisation of dural arteriovenous fistula via arterial and venous pathways: preliminary experience and evaluation of the short-term outcomes. Br J Radiol. 2012 Aug;85(1016):e395-403. doi: 10.1259/bjr/25192972. Epub 2012 Feb 28. PMID 22374275
- [Background] Maimon S, Nossek E, Strauss I, Blumenthal D, Frolov V, Ram Z. Transarterial treatment with Onyx of intracranial dural arteriovenous fistula with cortical drainage in 17 patients. AJNR Am J Neuroradiol. 2011 Dec;32(11):2180-4. doi: 10.3174/ajnr.A2728. Epub 2011 Oct 13. PMID 21998110
- [Background] van Rooij WJ, Sluzewski M. Curative embolization with Onyx of dural arteriovenous fistulas with cortical venous drainage. AJNR Am J Neuroradiol. 2010 Sep;31(8):1516-20. doi: 10.3174/ajnr.A2101. Epub 2010 Apr 15. PMID 20395390